CLINICAL TRIAL: NCT04857333
Title: Dynamic Evolution of Pulmonary Nodules and Influence Factors of Its Clinical Decision-making: A Prospective Cohort Study
Brief Title: Dynamic Evolution of Pulmonary Nodules and Influence Factors of Its Clinical Decision-making
Acronym: DEPICT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: GuiBin Qiao (Other)
Responsible Party: Sponsor-Investigator, GuiBin Qiao, Administrative Director, Department of Thoracic Surgery, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Other Study IDs: KY-Q-2021-005-03
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Nodule, Solitary; Pulmonary Nodule, Multiple
Keywords: Pulmonary nodule; Radiologic picture; Prospective observatory study; Psychological state; Decision-making
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules | interventions — Tomography, X-Ray Computed; Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Nodule: Patients are recommended for using antibiotics, solely follow-up or surgical resection according to the current clinical guideline for management of indeterminate pulmonary nodule. No intervention is administered for this observatory study.
  Interventions: Diagnostic Test: CT scan; Drug: Antibiotics; Procedure: Surgical Resection

INTERVENTIONS:
Diagnostic Test: CT scan — For patients with low-risk pulmonary nodules, follow-up CT scan is recommended
Drug: Antibiotics — For pulmonary nodules with features of infectious disease, antibiotics is recommended
Procedure: Surgical Resection — For persistent high-risk pulmonary nodules, surgical resection is recommended

SUMMARY:
The researchers are aimed to investigate the dynamic evolution of indeterminate pulmonary nodules by a long-term follow-up of patients with different characteristics. Influence factors of clinical decision-making that might contribute to overtreatment or delayed treatment will also be studied.

DETAILED DESCRIPTION:
This observatory study prospectively recruits patients with indeterminate pulmonary nodules identified in computed tomography (CT) scans from thoracic clinic. The radiological features and their chronological changes during follow-up period will be recorded in detail. Subgroup analyses will be performed based on the clinical and demographic characteristics of patients (including symptomatic information, comorbidities, family history, antibiotic usage, etc). Hospital Anxiety and Depression Scale (HADS) is collected from each patient at multiple time points to evaluate the patients' psychological status and its impact on clinical decision-making. The interaction analyses between individual characteristics (such as education level, occupation, disease cognitive level, etc) and Hospital Anxiety and Depression Scale will also be performed. The researchers aim to provide high-quality evidence for the formulation of a precise follow-up and management plan for patients with pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pulmonary nodules ≤ 3cm
2. Patients who provide electronic, written or oral consent to be enrolled in the follow-up cohort

Exclusion Criteria:

1. Patients with a surgical history of pulmonary nodules;
2. Patients who have obtained pathological diagnosis through surgery or non-surgical methods such as puncture;
3. Patients with pulmonary nodules that are likely metastatic from other sites;
4. Refuse to participate in this study.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All participants in this study are diagnosed with solitory or multiple indeterminate pulmonary nodules( ≤ 3cm ), and are willing to be followed-up for continous collection of their related disease information.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to surgical resection | The date of first documented diagnosis of pulmonary nodule by CT scan to the date of surgical resection, up to 60 months
  Time calculated from the date of identification of pulmonary nodule to the date of surgical resection
Time to progression | The date of first documented diagnosis of pulmonary nodule by CT scan to the date of documented progression by CT scan, up to 60 months
  Time calculated from the date of identification of pulmonary nodule to the date of progression of pulmonary nodule based on evaluation of CT imaging

SECONDARY OUTCOMES:
Proportion of malignancy | The date of first documented diagnosis of pulmonary nodule by CT scan to the date of surgical resection, up to 60 months
  Proportion of malignant findings by pathological examination in all patients receiving surgical resection
Change of Hospital Anxiety and Depression Scale-Anxiety (HADS-A) score | The date of enrollment in our cohort study when Hospital Anxiety and Depression Scale is measured to the date when primary endpoint( surgical resection) is reached, up to 60 months, with multiple measurements.
  The differences of Hospital Anxiety and Depression Scale-Anxiety (HADS-A) scores of the same patients before and after surgical resection. This 7-item checklist is a part of the Hospital Anxiety and Depression Scale, which is used for assessment for the status of anxiety. The maximal score for HADS-A is 21. Scores of greater than or equal to 11 on either scale indicate a definitive case. Scores of 0-7 are defined to be normal, while scores of 8-10 are defined to be borderline abnormal (borderline case).
Change of Hospital Anxiety and Depression Scale-Depression (HADS-D) score | The date of enrollment in our cohort study when Hospital Anxiety and Depression Scale is measured to the date when primary endpoint( surgical resection) is reached, up to 60 months, with multiple measurements.
  The differences of Hospital Anxiety and Depression Scale-Depression (HADS-D) scores of the same patients before and after surgical resection. This 7-item checklist is a part of the Hospital Anxiety and Depression Scale, which is used for assessment for the status of depression. The maximal score for HADS-D is 21. Scores of greater than or equal to 11 on either scale indicate a definitive case. Scores of 0-7 are defined to be normal, while scores of 8-10 are defined to be borderline abnormal (borderline case).

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
All individual participant data are strictly protected for patient privacy according to the agreement in Informed Consent Form.

REFERENCES:
- [Derived] Wu J, Zhuang W, Chen R, Xu H, Li Z, Lan Z, Xia X, He Z, Li S, Deng C, Xu W, Shi Q, Tang Y, Qiao G. Impact of surgery versus follow-up on psychological distress in patients with indeterminate pulmonary nodules: A prospective observational study. Qual Life Res. 2025 Apr;34(4):1167-1177. doi: 10.1007/s11136-024-03876-w. Epub 2025 Jan 15. PMID 39812961
- [Derived] Zhuang W, Tang Y, Xu W, Huang S, Deng C, Chen R, Zhang D, Zeng C, Tian D, Ben X, Lan Z, Wu H, Gao Z, Wang M, Chen Y, Shi Q, Qiao G. Should psychological distress be listed as a surgical indication for indeterminate pulmonary nodules: protocol for a prospective cohort study in real-world settings. J Thorac Dis. 2022 Mar;14(3):769-778. doi: 10.21037/jtd-21-1423. PMID 35399240